CLINICAL TRIAL: NCT03155269
Title: Impact of a Nutritional Supplement on Bone Turnover Markers in Indian Healthy Premenopausal Women (25-45 Yrs; Inclusive) After 6 Months of Intervention: a Randomised Double Blind Controlled Trial
Brief Title: To Investigate the Impact of a Nutritional Supplement on Bone Turnover Markers in Indian Healthy Premenopausal Women (25- 45 Years) After 6 Months of Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 207192
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-01

CONDITIONS: Growth and Development

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1- Protein rich beverage powder fortified with MMN (Experimental): Participants will be administered orally two doses of cereal based fortified beverage (30 grams powder made up in 200 milliliter (mL) water) daily in the morning and evening for 6 months.
  Interventions: Dietary Supplement: Fortified Beverage Powder
- Group 2 -Low protein non-fortified iso-caloric beverage powder (Other): Participants will be administered orally two doses (in morning and evening) of low protein non fortified isocaloric beverage (30 grams powder made up in 200 mL water) daily for 6 months.
  Interventions: Dietary Supplement: Non fortified beverage Powder

INTERVENTIONS:
Dietary Supplement: Fortified Beverage Powder — The tumbler will be filled with water up to the 200 mL mark. The entire contents of one sachet (Fortified beverage powder) will be gradually emptied in the tumbler with intermittent stirring to avoid formation of lumps. The reconstituted product will be consumed by the participants immediately orally.
  Arms: Group 1- Protein rich beverage powder fortified with MMN
Dietary Supplement: Non fortified beverage Powder — The tumbler will be filled with water up to the 200 mL mark. The entire contents of one sachet (Non fortified beverage powder) will be gradually emptied in the tumbler with intermittent stirring to avoid formation of lumps. The reconstituted product will be consumed by the participants immediately orally.
  Arms: Group 2 -Low protein non-fortified iso-caloric beverage powder

SUMMARY:
To investigate the effect of nutritional supplement on bone turnover markers (which are sensitive and respond quickly to nutrition or drug intervention) in Indian healthy premenopausal women after 6 months of intervention.

DETAILED DESCRIPTION:
This will be a double blind, single-center, randomized-controlled trial testing the effect of fortified beverage on bone turnover markers as compared to placebo control in 25-45 years old premenopausal women. The study will consist of two groups: Group 1 (Test) - Protein rich beverage powder fortified with MMN and Group 2 (control) - Low protein non-fortified iso-caloric beverage powder.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Female Participants.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon physical examination.
* BMI between 18.0-30 (kg/m2, Kilograms Per Meter Square) inclusive.
* Women who understand, willing, able and likely to comply with all study procedures and restrictions.

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study or Women who have a positive urine pregnancy test.
* Women who have attained physiological menopause defined as those who have not had a menstrual period for consecutive 12 months.
* Women who are breast-feeding.
* Current (within 14 days of the start of the study) or regular use of any prescription, over the counter (OTC), vitamin supplements herbal medicine unless the medication has been approved by the study physician.
* Treatment with bisphosphonates (any dose within the previous 2 years) or other medications known to affect bone (within the previous 6 months).
* History of metabolic bone disease.
* Any hormonal disorders or disturbances.
* Bone fracture in last 12 months.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Participant is lactose intolerant.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit.
* Previous participation in this study.
* Recent history (within the last 1 year) of alcohol or other substance abuse.
* More than 2 Units of alcohol per day
* Smokers
* Currently taking any other health food drinks/beverages or supplements (including nutritional supplements e.g. multivitamins and/or herbal supplements e.g. ginkgo) or has been on supplements within a month prior to study start.
* Women who used medication known to influence bone mass and the use of calcium, vitamin D, and multivitamin supplements on a regular basis were stopped 2 months before the onset of the trial.
* An employee of the sponsor or the study site or members of their immediate family.
* Ongoing conditions known to cause abnormalities of calcium metabolism or skeletal health, malabsorption syndromes (such as coeliac or Crohn's disease), hyperthyroidism, hyperparathyroidism, hypo- or hypercalcaemia, osteomalacia, Paget's disease, and diabetes.
* Fracture in the past 12 months.
* Known chronic kidney disease or alcoholism.
* Obesity women ( Body Mass Index, BMI>30) and Thinness i.e. BMI<18 kg/m2
* Severely anemic (Hemoglobin, Hb<8 g/dl, Grams Per Decilitre).
* Undertaking excessive exercise (>2 strenuous* exercise sessions per week)
* Contraceptive injections within the previous year.
* Known histories of surgeries such as bilateral oophrectomy (surgical removal of ovaries)
* Diagnosed hypogondal states such as Turner syndrome, Klinfelter syndrome, Kallman
* syndrome, anorexia nervosa, hypothalamic amenorrhea or hyperprolactinemia
* Hemotological disorders e.g. Hemophilia, Leukemia and lymphomas monoclonal multiple myeloma, sickle cell disease, Thalassemia etc.
* Rheumatological and autoimmune disorders such as ankylosing spondylitis, rheumatoid arthritis, systemic lupus etc.
* Miscellaneous conditions and diseases such as Human Immunodeficiency Virus/acquired immunodeficiency syndrome (HIV/AIDS), alcoholism, amyloidosis, chronic metabolic acidosis, Chronic Obstructive Pulmonary Disease (COPD), congestive heart failure, depression etc.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 114 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Pune, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in India.
Pre-assignment Details: A total of 117 participates were screened, out of which 114 participants were enrolled and allocated to a randomized treatment in the study (57 participants in each group), and 3 participants were not randomized due to withdrawl of consent.
Groups:
- Test Product: Participants received the protein rich beverage powder fortified with multi-micronutrients (MMN). The dose was prepared by dissolving 30 grams (g) of powder in 200 milli-liters (mL) of water which was consumed orally twice-daily; morning and preferably in the evening, for 6 months.
- Reference Product: Participants received the low protein non fortified isocaloric beverage powder. The dose was prepared by dissolving 30 grams (g) of powder in 200 milli-liters (mL) of water which was consumed orally twice-daily; morning and preferably in the evening, for 6 months.
Period: Overall Study
Arm/Group | Test Product | Reference Product
Started | 57 | 57
Completed | 52 | 50
Not Completed | 5 | 7
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population included all randomized participants who received at least 1 dose of study treatment. This population was based on the treatment the participant actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Product | Reference Product | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Continuous [Mean (Standard Deviation); unit: Years] — All randomized participants were included for baseline evaluation. Safety Population included all randomized participants who received at least 1 dose of study treatment. This population was based on the treatment the participant actually received.
  Years | 35.0 (4.41) | 34.2 (4.79) | 34.6 (4.60)
Sex: Female, Male [Count of Participants; unit: Participants] — All randomized participants were included for baseline evaluation. Safety Population included all randomized participants who received at least 1 dose of study treatment. This population was based on the treatment the participant actually received.
  Participants
    Female | 57 | 57 | 114
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — All randomized participants were included for baseline evaluation. Safety Population included all randomized participants who received at least 1 dose of study treatment. This population was based on the treatment the participant actually received.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 57 | 57 | 114
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Agr group [Number; unit: Participants] — All randomized participants were included for baseline evaluation. Safety Population included all randomized participants who received at least 1 dose of study treatment. This population was based on the treatment the participant actually received.
  Participants
    Age 25- <35 years | 26 | 27 | 53
    Age 35- <=45 years | 31 | 30 | 61
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — All randomized participants were included for baseline evaluation. Safety Population included all randomized participants who received at least 1 dose of study treatment. This population was based on the treatment the participant actually received.
  Centimeters (cm) | 152.8 (4.92) | 154.1 (5.27) | 153.4 (5.12)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Safety Population included all randomized participants who received at least 1 dose of study treatment. This population was based on the treatment the participant actually received.
  Kilograms (kg) | 57.5 (7.14) | 59.6 (8.52) | 58.5 (7.89)
Body Mass Index [Mean (Standard Deviation); unit: Kilograms per meter squares (kg/m^2)] — Safety Population included all randomized participants who received at least 1 dose of study treatment. This population was based on the treatment the participant actually received.
  Kilograms per meter squares (kg/m^2) | 24.7 (2.98) | 25.0 (2.84) | 24.8 (2.90)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Cross Linking C-telopeptide of Type 1 Collagen (s-CTX-1) at 6 Months
Description: s-CTX-1 is a bone resorption marker which is used to assess the bone health. After 6 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. CTX-1 serum was analysed using biochemical tests from the samples stored. Decreased s-CTX-1 is associated with improved bone health.
Time Frame: At baseline and at 6 months
Population: The Intent-to-Treat (ITT) population (n=102) was comprised of all randomized participants who received at least 1 dose of study treatment and had at least 1 post-baseline (post-treatment) primary efficacy evaluation. This population was based on the treatment to which the participant was randomized.
Measure: Mean (Standard Deviation); unit: Micrograms per litres (mcg/L)
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
Micrograms per litres (mcg/L)
  At Baseline | 0.4440 (0.11932) | 0.4410 (0.16213)
  At 6 months | 0.2828 (0.14218) | 0.3245 (0.16755)
  Change from baseline at 6 months | -0.1612 (0.15011) | -0.1165 (0.16574)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Other; p = 0.1324, ANCOVA — The setting of the two-sided significance level of 0.025 was used for the 2 co-primary endpoints to ensure that the overall significance level for the primary endpoint was less than or equal to 0.05; Analysis was performed using ANCOVA model with product group and strata as fixed effects, and the corresponding baseline value as covariate; Mean Difference (Final Values) = -0.0423, 97.5% CI 2-sided [-0.1057 to 0.0211] — Difference is test product minus reference product such that a negative difference favors the test product

2. Primary Outcome: Change From Baseline in the Ratio of Carboxylated (c-OC) to Under-carboxylated Osteocalcin (Uc-OC) at 6 Months
Description: c-OC/ uc-OC is considered as a surrogate marker of bone formation which is used to assess the bone health. After 6 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. c-OC/ uc-OC levels were analysed using biochemical tests from the samples stored. Increased c-OC/ uc-OC is associated with improved bone health.
Time Frame: At baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
Ratio
  At baseline | 1.208 (0.7573) | 1.138 (0.6747)
  At 6 months | 1.492 (0.6666) | 1.251 (0.4858)
  Change from baseline at 6 months | 0.284 (0.8961) | 0.113 (0.7160)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Other; p = 0.0469, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.229, 97.5% CI 2-sided [-0.030 to 0.489] — Difference is test product minus reference product such that a negative difference favors the test product

3. Secondary Outcome: Change From Baseline in Serum Cross Linking C-telopeptide of Type 1 Collagen (s-CTX-1) at 3 Months
Description: s-CTX-1 is a bone resorption marker which is used to assess the bone health. After 3 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. CTX-1 serum was analysed using biochemical tests from the samples stored. Decreased s-CTX-1 is associated with improved bone health.
Time Frame: At baseline and at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
mcg/L
  At baseline | 0.4440 (0.11932) | 0.4410 (0.16213)
  At 3 months | 0.2996 (0.15762) | 0.3302 (0.16693)
  Change from baseline at 3 months | -0.1444 (0.14563) | -0.1108 (0.13265)

4. Secondary Outcome: Change From Baseline in the Ratio of Carboxylated (c-OC) to Under-carboxylated Osteocalcin (Uc-OC) at 3 Months
Description: c-OC/ uc-OC is considered as a surrogate marker of bone formation which is used to assess the bone health. After 3 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. c-OC/ uc-OC levels were analysed using biochemical tests from the samples stored. Increased c-OC/ uc-OC is associated with improved bone health.
Time Frame: At baseline and at 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
Ratio
  At baseline | 1.208 (0.7573) | 1.138 (0.6747)
  At 3 months | 1.706 (1.2083) | 1.192 (0.8305)
  Change from baseline at 3 months | 0.498 (1.3043) | 0.054 (0.8868)

5. Secondary Outcome: Change From Baseline in Urinary Cross Linking C-telopeptide of Type 1 Collagen at 3 Months and 6 Months
Description: Urinary-CTX-1 is a bone resorption surrogate marker which is used to assess the bone health. After 3 months and 6 months of taking the allocated product, spot urinary sample were collected. CTX-1 urine levels were analysed using biochemical tests from the samples stored. Decreased urinary CTX-1 is associated with improved bone health.
Time Frame: At baseline, at 3 and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
mcg/L
  At baseline | 23.153 (17.3511) | 25.137 (22.8524)
  At 3 months: number analyzed (Participants) | 51 | 50
  At 3 months | 21.105 (16.8386) | 31.864 (27.5339)
  Change from baseline at 3 months: number analyzed (Participants) | 51 | 50
  Change from baseline at 3 months | -1.309 (20.8967) | 6.727 (22.7372)
  At 6 months | 16.318 (17.1383) | 18.708 (20.6598)
  Change from baseline at 6 months | -6.835 (22.1252) | -6.429 (27.9624)

6. Secondary Outcome: Change From Baseline in Serum N-terminal Telopeptide of Type 1 Collagen (s-NTX-1) at 3 Months and 6 Months
Description: NTX-1 is a bone resorption surrogate marker which is used to assess the bone health. After 3 months and 6 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. NTX-1 serum was analysed using biochemical tests from the samples stored. Decreased s-NTX-1 is associated with improved bone health. The unit of measurement is nanomole bone collagen equivalent (NM BCE).
Time Frame: At baseline, at 3 months and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: NM BCE
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
NM BCE
  At baseline | 11.64 (3.373) | 11.87 (3.093)
  At 3 months: number analyzed (Participants) | 52 | 48
  At 3 months | 10.68 (6.315) | 10.00 (5.720)
  Change from baseline at 3 months: number analyzed (Participants) | 52 | 48
  Change from baseline at 3 months | -0.97 (6.466) | -1.99 (5.861)
  At 6 months | 8.22 (3.146) | 9.38 (4.157)
  Change from baseline at 6 months | -3.43 (4.072) | -2.49 (4.296)

7. Secondary Outcome: Change From Baseline in Serum Procollagen Type 1 N-terminal Propeptide (s-P1NP) at 3 Months and 6 Months
Description: P1NP is a bone formation surrogate marker which is used to assess the bone health being the most abundant protein of bone matrix. After 3 months and 6 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. P1NP serum was analysed using biochemical tests from the samples stored. Increased s-P1NP is associated with improved bone health.
Time Frame: At baseline, at 3 months and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
mcg/L
  At baseline | 59.61 (22.044) | 58.70 (23.133)
  At 3 months: number analyzed (Participants) | 52 | 49
  At 3 months | 46.64 (17.982) | 54.22 (20.592)
  Change from baseline at 3 months: number analyzed (Participants) | 52 | 49
  Change from baseline at 3 months | -12.96 (15.929) | -4.85 (16.498)
  At 6 months | 43.86 (14.194) | 51.12 (22.586)
  Change from baseline at 6 months | -15.75 (18.272) | -7.58 (18.037)

8. Secondary Outcome: Change From Baseline in Bone Specific Alkaline Phosphatase (BSAP) at 3 Months and 6 Months
Description: BSAP is a bone formation surrogate marker which is used to assess the bone health. After 3 months and 6 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. BSAP serum was analysed using biochemical tests from the samples stored. Increased s-BSAP is associated with improved bone health.
Time Frame: At baseline, at 3 months and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
mcg/L
  At baseline | 11.071 (4.1076) | 10.774 (3.0623)
  At 3 months: number analyzed (Participants) | 51 | 50
  At 3 months | 9.441 (4.3417) | 10.188 (3.0810)
  Change from baseline at 3 months: number analyzed (Participants) | 51 | 50
  Change from baseline at 3 months | -1.649 (1.8695) | -0.586 (1.7019)
  At 6 months | 10.013 (3.3193) | 11.754 (3.3887)
  Change from baseline at 6 months | -1.058 (4.1670) | 0.980 (1.4648)

9. Secondary Outcome: Change From Baseline in Serum Parathyroid Hormone (s-PTH) at 3 Months and 6 Months
Description: PTH is used to compare calcium concentration status which defines the healthy bones. Intact PTH is the biologically active form and is secreted when the calcium level is low. After 3 months and 6 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. PTH serum was analysed using biochemical tests from the samples stored. Decreased s-PTH is associated with improved bone health.
Time Frame: At baseline, at 3 months and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Picomole per liter (pmol/L)
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
Picomole per liter (pmol/L)
  At baseline: number analyzed (Participants) | 52 | 49
  At baseline | 5.73 (2.875) | 5.35 (2.499)
  At 3 months: number analyzed (Participants) | 50 | 50
  At 3 months | 4.99 (3.394) | 5.75 (2.602)
  Change from baseline at 3 months: number analyzed (Participants) | 50 | 49
  Change from baseline at 3 months | -0.66 (2.798) | 0.34 (2.479)
  At 6 months: number analyzed (Participants) | 51 | 49
  At 6 months | 7.27 (3.429) | 8.09 (4.303)
  Change from baseline at 6 months: number analyzed (Participants) | 51 | 48
  Change from baseline at 6 months | 1.53 (3.126) | 2.69 (4.143)

10. Secondary Outcome: Change From Baseline in Urinary Calcium at 3 Months and 6 Months
Description: Urinary calcium is used to compare calcium concentration status which defines the healthy bones. After 3 months and 6 months of taking the allocated product, spot urinary sample were collected. Urinary calcium was analysed using biochemical tests from the samples stored. Decreased urinary calcium is associated with improved bone health.
Time Frame: At baseline, at 3 months and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimoles per moles (mmol/mol)
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
Millimoles per moles (mmol/mol)
  At baseline: number analyzed (Participants) | 50 | 49
  At baseline | 104.5 (78.26) | 104.0 (82.26)
  At 3 months: number analyzed (Participants) | 51 | 48
  At 3 months | 161.5 (142.60) | 116.9 (131.53)
  Change from baseline at 3 months: number analyzed (Participants) | 49 | 47
  Change from baseline at 3 months | 61.3 (126.75) | 16.4 (98.00)
  At 6 months: number analyzed (Participants) | 45 | 49
  At 6 months | 338.3 (440.08) | 549.7 (851.54)
  Change from baseline at 6 months: number analyzed (Participants) | 43 | 48
  Change from baseline at 6 months | 235.3 (451.33) | 448.9 (846.48)

11. Secondary Outcome: Change From Baseline in Serum Calcium at 3 Months and 6 Months
Description: Serum calcium is used to compare calcium concentration status which defines the healthy bones. After 3 months and 6 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. Serum calcium was analysed using biochemical tests from the samples stored. Increased serum calcium is associated with improved bone health.
Time Frame: At baseline, at 3 months and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
Millimoles per liter (mmol/L)
  At baseline | 2.299 (0.0629) | 2.296 (0.0703)
  At 3 months: number analyzed (Participants) | 49 | 49
  At 3 months | 2.266 (0.0778) | 2.258 (0.0862)
  Change from baseline at 3 months: number analyzed (Participants) | 49 | 49
  Change from baseline at 3 months | -0.038 (0.0854) | -0.037 (0.0825)
  At 6 months | 2.359 (0.0835) | 2.326 (0.0792)
  Change from baseline at 6 months | 0.060 (0.0873) | 0.030 (0.0821)

12. Secondary Outcome: Change From Baseline in Serum Phosphorus at 3 Months and 6 Months
Description: Serum phosphorus is a diagnostic marker for assessment of healthy bones. After 3 months and 6 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. Serum phosphorus was analysed using biochemical tests from the samples stored. Increased serum phosphorus is associated with improved bone health.
Time Frame: At baseline, at 3 months and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
mmol/L
  At baseline | 1.138 (0.1286) | 1.127 (0.1378)
  At 3 months: number analyzed (Participants) | 49 | 49
  At 3 months | 1.157 (0.1879) | 1.184 (0.1621)
  Change from baseline at 3 months: number analyzed (Participants) | 49 | 49
  Change from baseline at 3 months | 0.023 (0.1832) | 0.062 (0.1580)
  At 6 months | 1.127 (0.1493) | 1.123 (0.1810)
  Change from baseline at 6 months | -0.012 (0.1617) | -0.004 (0.1940)

13. Secondary Outcome: Change From Baseline in Total Alkaline Phosphatase (ALP) at 3 Months and 6 Months
Description: ALP is a diagnostic marker of which is used to assess bone mineral density for assessment of healthy bones. After 3 months and 6 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. Serum ALP was analysed using biochemical tests from the samples stored. Increased serum ALP is associated with improved bone health.
Time Frame: At baseline, at 3 months and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
Units per liter (U/L)
  At baseline | 68.6 (25.94) | 70.4 (18.38)
  At 3 months: number analyzed (Participants) | 49 | 49
  At 3 months | 63.3 (23.43) | 67.7 (17.65)
  Change from baseline at 3 months: number analyzed (Participants) | 49 | 49
  Change from baseline at 3 months | -5.9 (8.43) | -2.3 (8.77)
  At 6 months | 63.4 (20.26) | 70.2 (16.94)
  Change from baseline at 6 months | -5.1 (19.15) | -0.3 (9.44)

14. Secondary Outcome: Change From Baseline in Serum Vitamin D3 Using 25-hydroxycholecalciferol (25 OH D3) at 3 Months and 6 Months
Description: Serum vitamin-D3 is used to analyse the status of vitamin-D profile which is necessary for healthy bones. The marker used for analyzing serum vitamin-D3 was 25 OH D3. After 3 months and 6 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. Serum vitamin-D3 was analysed using biochemical tests from the samples stored. Increased serum vitamin-D3 is associated with improved bone health.
Time Frame: At baseline, at 3 months and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
nmol/L
  At baseline | 44.4 (36.78) | 42.2 (20.42)
  At 3 months: number analyzed (Participants) | 51 | 50
  At 3 months | 31.8 (20.45) | 41.2 (23.97)
  Change from baseline at 3 months: number analyzed (Participants) | 51 | 50
  Change from baseline at 3 months | -9.3 (14.60) | -1.0 (16.44)
  At 6 months | 30.5 (21.78) | 35.2 (25.02)
  Change from baseline at 6 months | -13.9 (27.51) | -7.0 (20.36)

15. Secondary Outcome: Change From Baseline in Serum Selenium (Se) at 3 Months and 6 Months
Description: Serum Se is used to assess the status of micronutrient profile necessary for healthy bones. After 3 months and 6 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. Serum Se was analysed using biochemical tests from the samples stored. Increased serum Se is associated with improved bone health.
Time Frame: At baseline, at 3 months and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micromole per liter (mcmol/L)
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
Micromole per liter (mcmol/L)
  At baseline: number analyzed (Participants) | 52 | 49
  At baseline | 1.350 (0.1702) | 1.305 (0.1791)
  At 3 months: number analyzed (Participants) | 51 | 50
  At 3 months | 1.293 (0.2153) | 1.245 (0.2875)
  Change from baseline at 3 months: number analyzed (Participants) | 51 | 49
  Change from baseline at 3 months | -0.055 (0.2447) | -0.076 (0.2464)
  At 6 months | 1.407 (0.2773) | 1.347 (0.2560)
  Change from baseline at 6 months: number analyzed (Participants) | 52 | 49
  Change from baseline at 6 months | 0.057 (2.738) | 0.031 (0.2705)

16. Secondary Outcome: Change From Baseline in Plasma Zinc (Zn) at 3 Months and 6 Months
Description: Plasma Zn is used to assess the status of micronutrient profile necessary for healthy bones. After 3 months and 6 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. Plasma Zn was analysed using biochemical tests from the samples stored. Increased plasma Zn is associated with improved bone health.
Time Frame: At baseline, at 3 months and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
mcmol/L
  At baseline: number analyzed (Participants) | 52 | 47
  At baseline | 10.75 (1.746) | 10.64 (2.071)
  At 3 months: number analyzed (Participants) | 52 | 49
  At 3 months | 10.28 (1.758) | 10.05 (1.540)
  Change from baseline at 3 months: number analyzed (Participants) | 52 | 46
  Change from baseline at 3 months | -0.47 (1.988) | -0.61 (2.234)
  At 6 months | 10.33 (1.324) | 10.00 (1.562)
  Change from baseline at 6 months: number analyzed (Participants) | 52 | 47
  Change from baseline at 6 months | -0.43 (2.066) | -0.60 (2.241)

17. Secondary Outcome: Change From Baseline in Serum Folic Acid (Folate) at 3 Months and 6 Months
Description: Serum folic acid (folate) is used to assess the status of micronutrient profile necessary for healthy bones. After 3 months and 6 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. Plasma Zn was analysed using biochemical tests from the samples stored. Increased serum folate is associated with improved bone health.
Time Frame: At baseline, at 3 months and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
nmol/L
  At baseline: number analyzed (Participants) | 52 | 49
  At baseline | 18.84 (13.570) | 39.74 (138.032)
  At 3 months: number analyzed (Participants) | 49 | 46
  At 3 months | 26.40 (25.768) | 15.09 (7.430)
  Change from baseline at 3 months: number analyzed (Participants) | 49 | 45
  Change from baseline at 3 months | 7.72 (27.996) | -27.05 (139.528)
  At 6 months: number analyzed (Participants) | 50 | 49
  At 6 months | 43.93 (135.047) | 16.27 (6.496)
  Change from baseline at 6 months: number analyzed (Participants) | 50 | 48
  Change from baseline at 6 months | 24.94 (137.118) | -23.82 (137.006)

18. Secondary Outcome: Change From Baseline in Plasma Vitamin-B6 at 3 Months and 6 Months
Description: Plasma vitamin-B6 is used to assess the status of micronutrient profile necessary for healthy bones. After 3 months and 6 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. Plasma vitamin-B6 was analysed using biochemical tests from the samples stored. Increased plasma vitamin-B6 is associated with improved bone health.
Time Frame: At baseline, at 3 months and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
nmol/L
  At baseline: number analyzed (Participants) | 51 | 50
  At baseline | 23.6 (16.11) | 22.4 (13.83)
  At 3 months: number analyzed (Participants) | 51 | 48
  At 3 months | 32.9 (22.59) | 22.4 (37.39)
  Change from baseline at 3 months: number analyzed (Participants) | 50 | 48
  Change from baseline at 3 months | 10.3 (25.75) | -0.5 (35.70)
  At 6 months | 32.6 (19.76) | 19.4 (12.08)
  Change from baseline at 6 months: number analyzed (Participants) | 51 | 50
  Change from baseline at 6 months | 8.9 (25.01) | -3.1 (10.96)

19. Secondary Outcome: Change From Baseline in Serum Vitamin-B12 at 3 Months and 6 Months
Description: Serum vitamin-B12 is used to assess the status of micronutrient profile necessary for healthy bones. After 3 months and 6 months of taking the allocated product, blood sample was collected under 12-hour fasting condition. Blood serum of whole blood collected from each participant was then isolated by the method of centrifugation. Serum vitamin-B12 was analysed using biochemical tests from the samples stored. Increased serum vitamin-B12 is associated with improved bone health.
Time Frame: At baseline, at 3 months and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 52 | 50
pmol/L
  At baseline | 177.1 (75.10) | 209.6 (140.28)
  At 3 months: number analyzed (Participants) | 51 | 49
  At 3 months | 212.5 (96.68) | 190.2 (76.99)
  Change from baseline at 3 months: number analyzed (Participants) | 51 | 49
  Change from baseline at 3 months | 33.8 (57.94) | -18.7 (126.96)
  At 6 months: number analyzed (Participants) | 51 | 50
  At 6 months | 227.4 (95.43) | 205.4 (91.70)
  Change from baseline at 6 months: number analyzed (Participants) | 51 | 50
  Change from baseline at 6 months | 50.1 (90.08) | -4.2 (135.21)

ADVERSE EVENTS:
Time Frame: 180 days +/- 7
Arm/Group | Test Product | Reference Product
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 19/57 | 19/57
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=57) | Reference Product (N=57)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood PTH increased (Investigations) | 2 (2) | 7 (7)
Urine calcium/ creatinine ratio increased (Investigations) | 3 (3) | 6 (6)
Vitamin-D deficiency (Metabolism and nutrition disorders) | 7 (7) | 2 (2)
Vitamin-B 12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hunger (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/69/NCT03155269/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT03155269/SAP_001.pdf